CLINICAL TRIAL: NCT06238245
Title: A Prospective, Single-Arm Clinical Study of Anti-thymocyte Globulin-based Conditioning Regimen Combined With Post-Transplantation Cyclophosphamide for GVHD Prevention in Allogeneic HSCT After PD-1 Blockade
Brief Title: Combination of ATG-based Conditioning Regimen and PTCy for GVHD Prevention in Allo-HSCT After PD-1 Blockade
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATGPTCY-PD1&GVHD2023V1.0
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Graft-versus-host Disease; Hematological Malignancies
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — Cyclophosphamide; Antilymphocyte Serum

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination of PTCy and ATG for GVHD prophylaxis (Experimental): ATG (anti-thymocyte globulin, rabbit; 5 mg/kg, day -5 to -2) was used in matched sibling donor-HSCT. ATG (1.5 mg/kg, day -5; 2.5 mg/kg, day -4; mathematical function was then exploited to determine the total targeted ATG dose on day -3 to -2 based on concentrations of active ATG on day -5 to -4) was used in both haploidentical donor-HSCT and unrelated donor-HSCT. Reduced-dose PTCy (two doses of 14.5 mg/kg Cy was given on days +3 and +4 post-HSCT) was used of GVHD prophylaxis.
  Interventions: Drug: Cyclophosphamid

INTERVENTIONS:
Drug: Cyclophosphamid — ATG (anti-thymocyte globulin, rabbit; 5 mg/kg, day -5 to -2) was used in matched sibling donor-HSCT. ATG (1.5 mg/kg, day -5; 2.5 mg/kg, day -4; mathematical function was then exploited to determine the total targeted ATG dose on day -3 to -2 based on concentrations of active ATG on day -5 to -4) was used in both haploidentical donor-HSCT and mismatched unrelated donor-HSCT. Reduced-dose PTCy (two doses of 14.5 mg/kg Cy was given on days +3 and +4 post-HSCT) was used of GVHD prophylaxis.
  Other Names: Anti-thymocyte globulin

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of anti-thymocyte globulin combined with PTCy (post-HSCT cyclophosphamide, PTCy) in preventing graft-versus-host disease (GVHD) in allo-HSCT patients after anti-PD-1(anti-programmed cell death protein 1) antibody treatment. In this study, patients with hematological malignancies who needed to receive allo-HSCT after PD-1 antibody treatment were selected as the research subjects. Fludarabine and Busulfan was used as the conditioning regimen, and the dose of ATG (anti-thymocyte globulin, ATG) combined with PTCy was used as the GVHD prevention regimen. The aim of this study is to reduce the incidence of Regimen-Related Toxicity and GVHD without affecting engraftment and relapse, thereby reducing non-relapse mortality and further improving the survival of patients.

DETAILED DESCRIPTION:
ATG (anti-thymocyte globulin, rabbit; 5 mg/kg, day -5 to -2) was used in matched sibling donor-HSCT. ATG (1.5 mg/kg, day -5; 2.5 mg/kg, day -4; mathematical function was then exploited to determine the total targeted ATG dose on day -3 to -2 based on concentrations of active ATG on day -5 to -4) was used in both haploidentical donor-HSCT and unrelated donor-HSCT. Reduced-dose PTCy regimen: two doses of 14.5 mg/kg Cy were given on days +3 and +4 post-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≥ 18 years old, regardless of gender;
* (2) patients with hematological malignancies (including lymphoma, leukemia, myelodysplastic syndrome, etc.) who had received at least one course of PD-1 antibody treatment;
* (3) patients with indications for allo-HSCT, available donors (including matched sibling donors, haploidentical donors and unrelated donors), and no contraindications for transplantation;
* (4) patients suitable for conventional Bu/Flu conditioning regimen;
* (5) no serious heart, liver, kidney, lung and other important organ diseases;
* (6) Eastern Cooperative Oncology Group (ECOG) performance status score 0-2;
* (7) Hematopoietic stem cell transplantation comorbidity index (HCT-CI) score was 0-3;
* (8) expected survival time of at least 12 weeks;
* (9) women who are not pregnant or breastfeeding;
* (10) voluntary participation in clinical research; They or their legal guardians were fully aware of the study and signed informed consent. Willing to follow and complete all trial procedures;

Exclusion Criteria:

* (1) pregnant or lactating women;
* (2) other serious conditions that may limit enrollment (e.g., advanced infection, etc.);
* (3) unable to understand and follow the study protocol or sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-02-28 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
acute graft-versus-host disease | 100 days
  Acute graft-versus-host disease severity is usually graded (grades 0-IV) by the pattern of organ involvement using the classic Glucksberg-Seattle criteria (GSC). Higher grades mean a worse outcome.

SECONDARY OUTCOMES:
chronic graft-versus-host disease | 1-year
  The National Institutes of Health scoring system (National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report) was used to define chronic GVHD. The standardization provided by the National Institutes of Health (NIH) 2005 and 2014 consensus projects has helped improve diagnostic accuracy and severity scoring (including grades mild, moderate, and severe) for clinical trials. Higher scores mean a worse outcome.
recurrence free survival | 1-year
  Recurrence Free Survival is defined as the time interval between the day of reference in the study (date of randomization, date of diagnosis, etc.) and the date of local relapse/recurrence or regional relapse/recurrence or death (all causes) whichever occurs first.
non-relapse mortality | 1-year
  Non-relapse mortality was defined as death from any cause other than malignancy relapse.
cumulative incidence of relapse | 1-year
  cumulative incidence of relapse was measured from the date of transplantation until the date of hematologic relapse.
overall survival | 1-year
  The time from transplantation to any cause death or the last follow-up was defined as overall survival.
GVHD-free/ relapse-free survival | 1-year
  GVHD-free/ relapse-free survival events were defined as grade 3-4 aGVHD or cGVHD requiring systemic immunosuppressive treatment, disease relapse, or any-cause death during the first 12 months after allogeneic HCT.
PD-L1 expression in acute myeloid leukemia bone marrow cells | Up to 1 year post-treatment
  The expression levels of PD-L1 in acute myeloid leukemia bone marrow cells will be assessed at the 28th day after each medication cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoning Gao, Doctor, Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Wang N, Wang L, Du J, Li F, Shao Y, Peng B, Luan S, Wang L, Jin X, Gao C, Dou L, Liu D. Targeted dosing of anti-thymocyte globulin in adult unmanipulated haploidentical peripheral blood stem cell transplantation: A single-arm, phase 2 trial. Am J Hematol. 2023 Nov;98(11):1732-1741. doi: 10.1002/ajh.27068. Epub 2023 Sep 14. PMID 37706580
- [Background] Gao XN, Su YF, Li MY, Jing Y, Wang J, Xu L, Zhang LL, Wang A, Wang YZ, Zheng X, Li YF, Liu DH. Single-center phase 2 study of PD-1 inhibitor combined with DNA hypomethylation agent + CAG regimen in patients with relapsed/refractory acute myeloid leukemia. Cancer Immunol Immunother. 2023 Aug;72(8):2769-2782. doi: 10.1007/s00262-023-03454-y. Epub 2023 May 11. PMID 37166484